CLINICAL TRIAL: NCT04020835
Title: Exploring Biopsychosocial Mechanisms of Abdominal Pain in Inflammatory Bowel Disease and Irritable Bowel Syndrome
Brief Title: Understanding Abdominal Pain in IBD and IBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 253660
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Abdominal Pain; Inflammatory Bowel Diseases; Irritable Bowel Syndrome
MeSH Terms: conditions — Abdominal Pain; Inflammatory Bowel Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — stool sample (faecal calprotectin)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abdominal pain is a central symptom of Inflammatory Bowel Disease (IBD) and Irritable Bowel Syndrome (IBS). IBD is an autoimmune disease characterized by inflammation of the gastrointestinal tract. IBS does not have clear biomarkers and is diagnosed based on symptom reports. The aim of this study is to explore biopsychosocial factors which may perpetuate and/or increase the severity of pain in these conditions. The main focus will be on the role of top-down brain processes in the experience of abdominal pain.

DETAILED DESCRIPTION:
It remains unclear why a large proportion of people with inflammatory bowel disease (IBD) report ongoing abdominal pain during remission or why people with irritable bowel syndrome (IBS) develop abdominal pain. One theory is that people with chronic pain have somehow grown more sensitive.

It is assumed that such heightened sensitivity depends both on bottom-up processing and top-down processing. Bottom-up processing refers to information that is relayed to the brain along so-called afferent fibres. Top-down processing refers to feedback provided by the brain to lower areas along efferent fibres.

The investigators will (1) measure the capacity of people to inhibit pain through top-down processing, (2) test if the human pain experience is enhanced due to sustained activation of certain afferents, and (3) assess to what extent people are impacted by psychosocial inhibition and activation factors. Results of people with IBS in remission will be compared with the results of two groups of people with IBD (those with pain and those without) and the investigators will explore if their measurements differentiate between groups.

It is hypothesized that (1) IBS patients and IBD patients with abdominal pain will be less able to inhibit their pain compared to IBD patients without abdominal pain (2) IBS patients and IBD patients with abdominal pain will score higher on psychosocial inhibition factors and lower on psychosocial activation factors when compared to IBD patients without abdominal pain. (3) In the total cohort, laboratory measures of pain inhibition will correlate with self-reported psychosocial inhibition and activation factors. (4) IBS patients and IBD patients with abdominal pain will show more temporal summation compared to IBD patients without abdominal pain.

ELIGIBILITY:
General inclusion criteria:

* Aged 18 and over
* Sufficient command of written and spoken English

IBD in remission inclusion criteria:

* Proof of diagnosis of IBD (Crohn's disease or ulcerative colitis) for more than 6 months - - Clear indicators of remission: on faecal calprotectin (≤200 µg/g) or measurements of C-reactive protein (CRP; ≤10 mg/dl) within the last 3 months or as part of recruitment
* No previous episodes of acute or sub-acute obstruction

IBS inclusion criteria:

* Current diagnosis of IBS measured with Rome IV criteria
* No serious other bowel diseases

Exclusion criteria:

* Major abdominal surgery in the last 6 months, or 3 or more previous major abdominal surgeries
* Pregnancy or childbirth in the last 6 months
* Any other diagnosed medical condition that may explain abdominal pain, including but not limited to known gynaecological conditions such as endometriosis and known post-surgical adhesions
* Any diagnosed co-morbid medical conditions associated with known neuropathy, such as diabetic neuropathy, renal neuropathy, multiple sclerosis
* Use of opioids in the last week
* Use of anti-depressants used as pain medication in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with quiescent Inflammatory Bowel Disease or Irritable Bowel Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficiency of inhibitory pain modulation, comparing patients with IBS or quiescent IBD | January 31, 2020
  Measured with Conditioned Pain Modulation test.
  Two inflatable pressure cuffs are secured around the caffs of subjects and then inflated. Pressure pain detection threshold (PDT) and pressure pain tolerance (PTT) are assessed on a subject's dominant leg. PDT is the first sensation of pain and PTT is defined as the point a subject no longer want the cuff to inflate. A VAS device allows participants to report their pain levels by moving a sliding button along a continuous line between two endpoints (0=no pain to 10=worst pain imaginable).
  After a second baseline measure on the non-dominant leg CPM is assessed: the cuff on the non-dominant leg is inflated to 70% of the subject's PTT, then after 15 seconds the cuff on the dominant leg is inflated. If pain modulation is achieved, the subject will show increased threshold and tolerance levels during CPM. The CPM-effect is defined as the difference between baseline and conditioning measurements of both PDT and PTT.
Contribution of socio-demographic, clinical and psychosocial factors to the efficiency of inhibitory pain modulation | January 31, 2020
  Measured with a range of questionnaires, i.e.: Brief Pain Inventory Short Form (BPI), painDETECT questionnaire, Patient Health Questionnaire-9, Generalized Anxiety Disorder-7, Visceral Sensitivity Index, Pain Catastrophising Scale, Cognitive and Behavioural Response to Symptoms Questionnaire, Pain Self Efficacy Questionnaire, Chronic Pain Acceptance Questionnaire-8, and Mental Health Continuum Short-Form

SECONDARY OUTCOMES:
Pain facilitation, comparing patients with IBS and quiescent IBD | January 31, 2020
  Measured with Temporal Summation (TS) test.
  TS will be carried out on the dominant leg dominant. A series of 10 rapid stimuli will be given at a rate of 0.5 Hz (1-second of pressure at 1-second intervals). The cuff pressure-level of the stimuli will be determined by the pressure pain tolerance level of the subject. In each instance the subject will rate the painfulness of the stimulus using the VAS. The VAS rating for each stimulus will be relative to the painfulness of the previous stimulus in the train of stimuli, i.e. the subject does not return the VAS scale to zero after each stimulation. In other words, if the painfulness of a stimulus is more intense than the previous stimulus, the VAS scale is increased. If the painfulness of stimulus is less intense than the previous stimulus, the VAS scale is decreased. If the sensation remains the same between stimuli, then the VAS scale is not changed.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London